CLINICAL TRIAL: NCT00657163
Title: Effects of 3 Months Daily Treatment With Selective Serotonin Reuptake Inhibitor (SSRI, Fluoxetine) on Motor Rehabilitation After Ischemic Stroke. FLAME Trial
Brief Title: Fluoxetine on Motor Rehabilitation After Ischemic Stroke
Acronym: FLAME
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0300501; French PHRC
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Last update posted 2011-09-16 (Estimated); Status verified 2009-07

CONDITIONS: Ischemic Stroke; Motor Impairment
Keywords: Stroke recovery; Pharmacological modulation; Selective Serotonin Reuptake Inhibitor (SSRI); Fluoxetine; Brain plasticity; Ischemic Stroke and Motor impairment; Modulation of recovery and cerebral plasticity by Fluoxetine
MeSH Terms: conditions — Ischemic Stroke | interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): fluoxetine
  Interventions: Drug: fluoxetine
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: fluoxetine — fluoxetine per os 20 mg daily
  Other Names: PROZAC
  Arms: 1
Drug: placebo — placebo per os daily
  Arms: 2

SUMMARY:
Recovery from stroke is a major process and, except for acute intravenous thrombolysis, no treatment able to enhance recovery has yet been validated. Some drugs may have a positive effect when combined with physical rehabilitation. Previous studies have shown a potential effect of catecholaminergic drugs on cerebral plasticity of stroke patients. In 2001, our group has demonstrated in a small group of stroke patients (n=8) that a single dose of fluoxetine (Selective Serotonin Reuptake Inhibitor - SSRI) improved motor performance and modulated cerebral plasticity. We conducted a phase IIb prospective, double-blind, randomized, placebo controlled study to assess the effect of a daily treatment with fluoxetin (20 mg) on motor performance in patients with mild to severe motor deficit after ischemic stroke.

DETAILED DESCRIPTION:
We project to include in the study a maximum of 168 patients with a recent (5 to 10 days) ischemic stroke and unilateral motor deficit in order to obtain 100 completed patients. Nine stroke centers in France are involved.

Each patient will receive daily, during three months, 20 mg of fluoxetin or placebo.

Patients will be evaluated at inclusion, day 30, M3 (3 months), M12.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged from 18 to 85
* No motor relapse from a previous stroke
* Inclusion from day 5 to day 10 after stroke
* Ischemic stroke with unilateral motor deficit
* Motor NIHSS ≥ 5 on the affected side of the body
* NIHSS < 20
* Fugl Meyer Motor Scale <55
* Modified Rankin Scale between 1 and 5
* Informed consent obtained from the subject or a member of his family

Exclusion Criteria:

* Pregnant or breast-feeding woman
* Woman able to procreate without valid contraception
* Subject protected by law
* Concomitant disease with unfavourable prognosis within 1 year
* Drug addiction
* Allergy to fluoxetine
* Hepatic failure (TGO and TGP >2N)
* Permanent Renal failure (Creatinin >180micromol/l)
* Patients treated by tricyclic antidepressant, selective serotonin reuptake inhibitor, monoamine oxidase inhibitor (IMAO), and neuroleptics in the past month
* Depression requiring pharmacological treatment
* Previous stroke with motor relapse
* Fugl Meyer Motor Scale > 55
* Modified Rankin Scale = 0 or 6
* Patients needing carotid surgery within 3 months
* Aphasia preventing correct evaluation of motor and depression scales.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Progression in the Fugl-Meyer Motor Scale | M3 (3 months)

SECONDARY OUTCOMES:
Fugl-Meyer Stroke Scale | M12 (12 months)
NIH stroke scale | M3 and M12
MADRS depression scale | M3 and M12
Modified Rankin scale | M3 and M12
Mortality | M3 and M12

CONTACTS AND LOCATIONS:
Overall Officials: François Chollet, PhD, Principal Investigator — University Hospital, Toulouse
Locations (9):
- France (9):
  - University Hospital, Besançon
  - University Hospital René Dubos, Cergy-Pontoise
  - University Hospital, Dijon
  - University Hospital, Grenoble
  - University Hospital, Nantes
  - University Hospital Pitié Salpétrière, Paris
  - University Hospital Sainte Anne, Paris
  - University Hospital Rangueil, Toulouse
  - University Hospital Purpan, Toulouse

REFERENCES:
- [Background] Pariente J, Loubinoux I, Carel C, Albucher JF, Leger A, Manelfe C, Rascol O, Chollet F. Fluoxetine modulates motor performance and cerebral activation of patients recovering from stroke. Ann Neurol. 2001 Dec;50(6):718-29. doi: 10.1002/ana.1257. PMID 11761469
- [Background] Dam M, Tonin P, De Boni A, Pizzolato G, Casson S, Ermani M, Freo U, Piron L, Battistin L. Effects of fluoxetine and maprotiline on functional recovery in poststroke hemiplegic patients undergoing rehabilitation therapy. Stroke. 1996 Jul;27(7):1211-4. doi: 10.1161/01.str.27.7.1211. PMID 8685930
- [Derived] Chollet F, Tardy J, Albucher JF, Thalamas C, Berard E, Lamy C, Bejot Y, Deltour S, Jaillard A, Niclot P, Guillon B, Moulin T, Marque P, Pariente J, Arnaud C, Loubinoux I. Fluoxetine for motor recovery after acute ischaemic stroke (FLAME): a randomised placebo-controlled trial. Lancet Neurol. 2011 Feb;10(2):123-30. doi: 10.1016/S1474-4422(10)70314-8. Epub 2011 Jan 7. PMID 21216670